CLINICAL TRIAL: NCT04471389
Title: Effect of the Interaction Between Environmental Factors and Salt-sensitive Genomics on Long-term Blood Pressure in Chinese Population
Brief Title: Longitudinal Follow-up Study in Two Chinese Hypertension Cohorts
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2019-004
Record Dates: First submitted 2020-06-21; First posted 2020-07-15 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Hypertension
Keywords: blood pressure; Salt-sensitive; Left Ventricular Hypertrophy; Vascular Stiffness; Carotid Artery Diseases
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular; Carotid Artery Diseases | interventions — Incidence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Meixian county adult salt-sensitive hypertension study is a family-based dietary interventional study. Whole blood specimen was collected from each participant who underwent a chronic salt load and potassium supplementation trial. Genomic DNA was extracted from whole blood specimen using the GOLDMAG Whole Blood Genomic DNA Purification Kit.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hanzhong adolescent hypertension cohort: A total of 4623 adolescents aged 6-15 years old in Hanzhong rural areas was recruited in 1987. During the follow-up period, the information about the incidence and risk factors of hypertension will be collected.
  Interventions: Other: Incidence and risk factors of hypertension
- Mei county adult salt-sensitive hypertension cohort: A total of 675 individuals from 126 families were recruited in this family-based dietary intervention study. A community-based BP screening was conducted among adults aged 18-60 years in the study villages. The probands who had a mean systolic BP (SBP) between 130-160 mmHg and/or a diastolic BP (DBP) between 85-100 mmHg and no use of antihypertensive medications and their parents, siblings, spouses, and offspring were recruited in this study. During the follow-up period, the information about the incidence and risk factors of hypertension will be collected.
  Interventions: Other: Incidence and risk factors of hypertension

INTERVENTIONS:
Other: Incidence and risk factors of hypertension — During the follow-up period, General information(age, sex, BMI, blood pressure, the history of drink and smoke, medical history, etc). Blood biochemistry parameters（Lipid, hsCRP levels, etc）and other laboratory examination parameters(arterial stiffness, IMT, FMD) will be collected.

SUMMARY:
Essential hypertension is a complex trait that results from interaction between environmental factors and genetic factors. Salt sensitivity is the genetic susceptibility of blood pressure to salt, and it is an intermediate genetic phenotype of essential hypertension. This study aims to investigate the effects of interaction between salt sensitivity genomics and environmental factors on long-term blood pressure (BP) and target organ damage based on two established cohorts including "the cohort of Hanzhong adolescent hypertension study" and "the cohort of Mei county adult salt-sensitive hypertension study". Firstly, the Hanzhong cohort-based follow-up study is designed to observe the track of BP from childhood, and to explore the effects of many risk factors (such as salt-sensitivity, obesity et al) on long-term BP changes and the occurrence of TODs. In addition, by using DNA samples collected from subjects of "Mei county adult salt-sensitive hypertension study" in which all participants had completed a chronic salt loading and potassium intervention trial, investigators attempt to carry out whole-exome sequencing (WES), whole-genome DNA methylation and transcriptome detection, and analyze the relationship between salt sensitivity genomics and BP responses to dietary sodium/potassium intervention, long-term BP change, the risk of target organ damages. Investigators aim to explore the role of risk factors, including salt sensitivity, in the development of hypertension, and to illustrate the effects of interaction between salt sensitivity genomics and environmental factors on hypertension and target organ damage. This study would enable the investigators to further explore the genetic mechanism of essential hypertension, to identify new genetic markers for predicting early hypertension and target organ damage as well as to provide the basis for the prevention, targeted treatment, and new drugs development of hypertension in the future.

DETAILED DESCRIPTION:
This study is a longitudinal cohort follow-up study. The main contents include:

(1) Questionnaire design: the questionnaire is designed according to the research contents and purposes. The standard questionnaires will be used to collect the general information, dietary habits, lifestyle, medical history, and family history etc. (2) Anthropometric measurements: blood pressure, pulse, height, body weight, waist and hip circumference will be acquired by medical practitioners who received professional training based on World Health Organization (WHO) standards, and passed relevant examinations. (3) Blood and urine samples collection: morning fasting blood, nocturia, and 24-hour urine specimen will be collected by medical staffs, and blind tubes will be set up according to 5% of the total samples. Blood biochemistries including serum total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, fasting glucose, creatinine and hsCRP can be measured using automatic biochemical analyzer. The sodium and potassium concentrations in the urine will be measured by flame photometry. The total sodium and potassium excretions in urine in 24h were calculated by multiplying the concentration and 24-h volume of urine. (4) Auxiliary examinations: Auxiliary examinations including carotid intima-media thickness, endothelium-dependent vasodilation (FMD), measurements of brachial-ankle pulse wave velocity (baPWV) and electrocardiographic parameters. The measurement will be done in hospitals by medical practitioners who received professional trainings and passed relevant examinations. (5) Whole-exome sequencing: Genomic DNA will be isolated from blood samples and subjected to exome capture, followed by next-generation sequencing on the Roche NimbleGen system. (6) Whole-genome DNA methylation analysis: levels of DNA methylation will be quantified using the Illumina Infinium HumanMethylation450K Beadchip array (HM450K). (7) Transcriptome sequencing: cDNA libraries will be sequenced via the Illumina HiSeqTM 2500 platform. (8) Data processing and statistics: investigators should input the data to the database, and utilize software such as Access, SPSS, STATA, CASAVA, MutSigCV, and Genome MuSic to analyze. (9) Quality control: ① Questionnaire is strictly designed and amended by epidemiologists and clinical experts. ② A standardized "Investigator Handbook" will be stipulated according to the guidelines. ③ Staff members are required to do a rigorous training and pass the exam. ④ The investigation process will be strictly supervised by the principal investigator. ⑤ Data entry uses the parallel double-entry method. ⑥ During laboratory testing, blank control and blind detection are applied to ensure the quality. ⑦ Data analysis is performed by 2-3 postgraduates, inconsistent data need to be double-checked.

ELIGIBILITY:
Inclusion Criteria:

1. Hanzhong cohort of Adolescent Hypertension Study:

   • adolescents aged 6-15 years old in over 20 schools of three towns (Qili, Laojun and Shayan) in Hanzhong, Shaanxi, China.
2. Mei county cohort of adult salt-sensitive hypertension study:

   * Han individuals in rural northern China
   * adults aged 18-60 years
   * individuals who had a mean systolic BP (SBP) between 130-160 mmHg and/or a diastolic BP (DBP) between 85-100 mmHg and no use of antihypertensive medications were identified as the proband
   * the probands'parents, siblings, spouses, and offspring were recruited for the study.

Exclusion Criteria:

* Secondary hypertension
* a history of severe cardiovascular disease
* chronic kidney disease or liver disease
* unable to complete the examination
* unable/refuse to sign the informed consent form

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: In March and April 1987, investigators established the cohort of Hanzhong Adolescent Hypertension Study. A total of 4,623 adolescents aged 6-15 years old in over 20 schools of three towns (Qili, Laojun and Shayan) in Hanzhong, Shaanxi, China were recruited. In 2003-2004, investigators established the cohort of Mei county adult salt-sensitive hypertension Study. This study was a family-based dietary intervention study conducted in a Han Chinese population from rural areas of northern China. A total of 675 subjects from 126 families were recruited in this cohort.
Sampling Method: Probability Sample
Enrollment: 5611 (Estimated)
Dates: Start 2021-09 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
blood pressure value(mmHg) | First day of the three-day follow-up period
  The follow-up study of these two cohorts will last approximately 24 months (Jan 2020 to Dec 2021). During this period, each subject will receive a three-day follow-up examination. Three BP (mmHg) measurements will be obtained using a mercury sphygmomanometer on the first day of the three-day follow-up period.

SECONDARY OUTCOMES:
Left ventricular hypertrophy (g/m^2) | During the three-day follow-up period
  The follow-up study of these two cohorts will last approximately 24 months (Jan 2020 to Dec 2021). During this period, each subject will receive a three-day follow-up examination. Left ventricular mass index (LVMI,g/m^2)will be measured using echocardiography during the three-day follow-up period.
Increased arterial stiffness (mm/s) | During the three-day follow-up period
  The follow-up study of these two cohorts will last approximately 24 months (Jan 2020 to Dec 2021). During this period, each subject will receive a three-day follow-up examination. Brachial-ankle pulse wave velocity (baPWV, mm/s) will be measured with Noninvasive automatic waveform analyzer during the three-day follow-up period.
Carotid artery wall thickening (mm) | During the three-day follow-up period
  The follow-up study of these two cohorts will last approximately 24 months (Jan 2020 to Dec 2021). During this period, each subject will receive a three-day follow-up examination. Carotid Intima media thickness (IMT, mm) will be measured using Color Doppler Ultrasound Diagnostic System during the three-day follow-up period.
Microalbuminuria (mg/24h) | Second day of the three-day follow-up period
  The follow-up study of these two cohorts will last approximately 24 months (Jan 2020 to Dec 2021). During this period, each subject will receive a three-day follow-up examination. On the second day, 24-hour urinary will be collected and the concentrations of microalbuminuria in the urine sample will be measured with Hitachi biochemical analyzer. The 24-hour microalbuminuria(mg/24h) of each subject is calculated as the concentration of microalbuminuria multiplied by the 24-hour urine volume of each individual.
whole exome sequencing | the whole year after the follow-up period
  After the two-year follow-up, sample examination and data analysis will take 12 months (Jan 2022 to Dec 2022). During this period, whole exome sequencing will be carried out on each sample using Illumina Hiseq 2500.
whole genome DNA methylation detection | the whole year after the follow-up period
  After the two-year follow-up, sample examination and data analysis will take 12 months (Jan 2022 to Dec 2022). During this period, whole genome DNA methylation detection will be carried out on each sample using illulIlina Human Melylation 450K Beadchip.
whole-genome transcriptome sequencing | the whole year after the follow-up period
  After the two-year follow-up, sample examination and data analysis will take 12 months (Jan 2022 to Dec 2022). During this period, whole-genome transcriptome detection will be carried out on each sample using Illumina HiseqTM 2500.

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Mu, doctor, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
The achievements will be evaluated by papers published in specialized journals with a peer-reviewed system, and the original dates can be disclosed according to requirements.

REFERENCES:
- [Result] Zheng W, Mu J, Chu C, Hu J, Yan Y, Ma Q, Lv Y, Xu X, Wang K, Wang Y, Deng Y, Yan B, Yang R, Yang J, Ren Y, Yuan Z. Association of Blood Pressure Trajectories in Early Life with Subclinical Renal Damage in Middle Age. J Am Soc Nephrol. 2018 Dec;29(12):2835-2846. doi: 10.1681/ASN.2018030263. Epub 2018 Nov 12. PMID 30420422
- [Result] Fang Y, Mu JJ, He LC, Wang SC, Liu ZQ. Salt loading on plasma asymmetrical dimethylarginine and the protective role of potassium supplement in normotensive salt-sensitive asians. Hypertension. 2006 Oct;48(4):724-9. doi: 10.1161/01.HYP.0000238159.19614.ce. Epub 2006 Sep 11. PMID 16966580